CLINICAL TRIAL: NCT07383077
Title: proTmedula- Temporal Profile of Potential Molecular Determinants of Spinal Cord Injury Rehabilitation and Regeneration
Brief Title: Molecular Determinants of Spinal Cord Injury Rehabilitation
Acronym: proTmedula
Status: Completed | Type: Observational
Sponsor: Prof. Sandra Vieira (Other)
Collaborators: Aveiro Institute of Biomedicine (iBiMED) (Unknown); Department of Medical Sciences, University of Aveiro (Unknown); Centro de Reabilitacao do Norte (Other); Unidade Local de Saude de Gaia e Espinho EPE (Other); Centro Academico Clínico Egas Moniz Health Alliance (Other)
Responsible Party: Sponsor-Investigator, Prof. Sandra Vieira, Prof. Sandra I. Vieira, Aveiro University
Organization: Aveiro University (Other)
Other Study IDs: ProTmedula 246/2019-2 SAcu-Chr; NCT06892106 ClinicalTrials.gov (Other: ClinicalTrials.gov)
Record Dates: First submitted 2026-01-17; First posted 2026-02-03 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Spinal Cord Injury
Keywords: Spinal Cord Injury; Rehabilitation; Regeneration; Omics; Biomarkers; Therapeutic targets; Translational
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, urine and fecal samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- SCI cohort: Spinal cord injury patients admitted for hospitalization at Centro de Reabilitação do Norte, Unidade Local de Saúde de Gaia e Espinho, E.P.E. categorized into two subgroups: with A or B (motor complete injuries) classification, or with C or D (motor incomplete) classification in The American Spinal Injury Association (ASIA) Impairment Scale (AIS).
- Able-bodied controls: Age, sex and body mass index-matched control group of participants recruited among able-bodied personnel from Centro de Reabilitação do Norte, Unidade Local de Saúde de Gaia e Espinho, E.P.E. or their relatives, without any known CNS disease.

SUMMARY:
This study main aim is to identify molecular determinants of better recovery following spinal cord injury (SCI), as biomarkers of neurological and/or functional improvement and a proxy for neuroregeneration. For that, omics analyses of several biological samples will be performed, to comprehensively portray the molecular and cellular profiles of the patients with SCI at key time points of the pathology: pre-rehabilitation, post-rehabilitation and one-year post-injury. The main question it aims to answer is: 'Are there specific molecules (and related biological pathways) that impact the functional recovery of spinal cord injury patients during the subacute phase, in a way that future targeted pharmacological or genetic interventions may improve SCI outcomes?'.

DETAILED DESCRIPTION:
BACKGROUND:

Spinal cord injury (SCI) is a devastating condition with no effective cure, that hinders motor, sensory and autonomic functions. Besides affecting the spinal cord parenchyma, SCI has various systemic impacts including altered metabolic states, chronic inflammation, gastrointestinal alterations like gut dysbiosis, and urinary dysfunctions. Given these systemic pathophysiological effects, and the physiological drainage of molecules from the cerebrospinal fluid into the bloodstream, SCI biomarkers may also be identified in the blood/serum, urine and feces.

This study hypothesizes that alterations in proteins, metabolites and gut bacteria from blood/serum, urine and/or feces, reflect and influence neurological and/or functional recovery of SCI patients. Thus, using high-throughput omics analyses, the investigators here aim to identify molecular determinants and microbiota taxa that correlate with clinical recovery measures (the motor scores assessed by the International Standards for Neurological Classification of Spinal Cord Injury - ISNCSCI, the American Spinal Injury Association (ASIA) Impairment Scale - AIS grades, the Spinal Cord Independence Measure - SCIM-IV, and the Functional Independence Measure - FIM). In parallel, the investigators also aim to monitor potential neuroregeneration-associated molecules identified in pre-clinical studies led by the investigators, such as project GoBack (New therapeutic targets for spinal cord injury regeneration - PTDC/CVT-CVT/32261/2017), project pAGE (Protein aggregation across the lifespan - CENTRO-01-0145-FEDER-000003), project MEDISIS (CENTRO-01-0246-FEDER-000018), and project ReConnect (Developing innovative therapies for spinal cord injury - COMPETE2030-FEDER-00891600).

STUDY OBJECTIVES:

This research work has the following main objectives:

1. To perform broad-spectrum omics analyses, including metabolomics, proteomics, microbiome, in samples from patients with SCI at different phases post-injury, including pre- and post-rehabilitation;
2. Correlate the levels of relevant molecules and microbiota taxa identified in the omics analyses with relevant clinical data (including vital data and outcome measures like AIS grades, ISNCSCI motor scores, and functional scales SCIM-IV and FIM), in a Systems Medicine approach to SCI;
3. To monitor potential biomarkers of spinal cord injury and neuroregeneration, discovered within the scope of the investigators' previous and ongoing pre-clinical projects in cell and animal models of SCI, and search for associations between these molecules and relevant clinical data.

EXPLORATORY OBJECTIVE:

To identify biomarkers that may help in prognosis, stratification and pharmacological adjustments, and/or serve as therapeutic targets, with the main aim to improve the quality of life of spinal cord injury patients, particularly by improving their functional competences and attenuate commorbidities.

STUDY DESIGN AND METHODOLOGY:

Observational, longitudinal, prospective cohort study involving 66 patients with subacute SCI (28 patients with A and B classification in ASIA Impairment Scale - AIS and 38 patients with C and D classification in AIS) and 40 able-bodied control participants, recruited from familiars, hospital personnel and the community.

PARTICIPANT RECRUITMENT:

Participants were recruited when admitted for hospitalization at the rehabilitation center "Centro de Reabilitação do Norte (CRN, ULSGE)". Inclusion and exclusion criteria were clearly defined to ensure a homogenous and representative study population.

DATA COLLECTION:

Clinical data, including neurological assessments (e.g., ASIA Impairment Scale), functional outcome measures (e.g. SCIM, FIM), and demographic information, were collected at three time points (T): T1: Admission to the rehabilitation unit (subacute phase, around 2 months post-injury). T2: Discharge from the rehabilitation unit (around 4 months post-injury). T3: One-year post-injury follow-up. Biological samples (blood, feces, and urine) were collected at each time point (T1, T2, and T3). The same biological samples were collected from controls at a single time point.

LABORATORY ANALYSES:

Metabolomics and Lipidomics analyses: Serum samples were analysed by Attenuated Total Reflection Fourier-Transform Infrared (ATR-FTIR) spectroscopy, fecal and serum samples by Nuclear Magnetic Resonance (NMR); serum samples will be analysed by Mass-spectrometry-based lipidomics.

Microbiome Analysis: Fecal samples undergone 16S rRNA gene sequencing to determine gut microbiota composition and diversity.

Immune Biomarker Quantification: Serum samples were analyzed by citometry multiplex array.

Proteomic analyses: Serum samples were analysed by Mass-spectrometry.

STATISTICAL ANALYSES:

Descriptive statistics (mean/median) were calculated for all outcome measures. Data association studies will be performed between molecular data (levels of microbiota taxa and/or molecules at a given time point, or their variation between time points) and continuous (e.g. ISNCSCI motor scores; SCIM-IV and FIM scores) and categorical clinical data (e.g. stratification by severity using AIS grades; medication intake).

Potential confounders (age, gender, injury level, time post-injury, etc.) and biases are being accounted for. Independent group comparisons (e.g., T1 cytokine levels) used t-tests or Mann-Whitney U-tests, while dependent group comparisons (e.g., cytokine changes within AIS groups) used paired t-tests or Wilcoxon tests. ANOVA, multivariate analyses, and generalized linear models (regression, mixed-model repeated measures) assessed inter-group data and associations between omics datasets and clinical measures. Multiomics analyses will be performed using prediction models.

ELIGIBILITY:
Inclusion Criteria:

* Clinically diagnosed with traumatic spinal cord injury
* Adults (≥18 years).
* Injury occurred less than 6 months ago (subacute phase).
* Classification A-D in The American Spinal Injury Association (ASIA) Impairment Scale (AIS).
* Any neurological level of injury.

Exclusion Criteria:

* Use of probiotics one-month prior admission.
* Use of immunomodulatory drugs one-month prior admission.
* Major gastrointestinal surgery in the last five years.
* Active gastrointestinal diseases.
* Other CNS diseases (besides SCI).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the North Rehabilitation Center ("Centro de Reabilitação do Norte, CRN-ULSGE") between 1st of May 2021 and 16th of October 2023, following a traumatic spinal cord injury.
Sampling Method: Non-Probability Sample
Enrollment: 106 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2023-10-16 (Actual); Study Completion 2023-10-16 (Actual)

PRIMARY OUTCOMES:
Molecular/cellular candidate biomarkers with a strong association to functional independence | From admission into the rehabilitation hospital (~2 months post-injury) until discharge (~4 months post-injury)
  Association between functional independence, assessed by the Spinal Cord Independence Measure, 4th version (SCIM IV), and by the Functional Independence Measure (FIM), with levels of specific molecular or cellular candidate biomarkers.
  Association studies will consider functional independence measures (at admission, their variation, and/or at discharge) and specific molecular or cellular candidate biomarkers, such as protein or bacterial levels (at admission, their variation, and/or at discharge).
Molecular/cellular candidate biomarkers with a strong association to neuromotor impairment | From admission into the rehabilitation hospital (~2 months post-injury) until discharge (~4 months post-injury)
  Association between total motor scores, assessed by the International Standards for Neurological Classification of Spinal Cord Injury (ISNCSCI), with levels of specific molecular or cellular candidate biomarkers.
  Association studies will consider ISNCSCI motor scores (at admission, their variation, and/or at discharge) and specific molecular or cellular candidate biomarkers, such as protein or bacterial levels (at admission, their variation, and/or at discharge).

SECONDARY OUTCOMES:
Molecular/cellular candidate biomarkers identified in the primary outcome measures with a strong association to neurological impairment | From admission into the rehabilitation hospital (~2 months post-injury), across discharge (~4 months post-injury), and until follow-up (1-year post-injury)
  Association between the grade determined by the American Spinal Injury Association (ASIA) Impairment Scale (AIS), with levels of molecular or cellular candidate biomarkers identified in the primary outcome measures.
  Association studies will consider AIS grades (at admission, at discharge, at one-year follow-up, and/or their variation between two time points) and previously identified molecular or cellular candidate biomarkers, such as protein or bacterial levels (at admission, at discharge, at one-year follow-up, and/or their variation between two time points).
Longitudinal profiles of key molecules (and bacteria) across post-intensive inpatient rehabilitation, and a period post-discharge (subacute and chronic phases) | From admission into the rehabilitation hospital (~2 months post-injury), across discharge (~4 months post-injury), and until follow-up (1-year post-injury)
  Relevant candidate biomarkers, identified in pre-clinical studies, or in targeted or omics analyses of this cohort's biological samples, measured through relative abundances or absolute concentrations, as determined by omics software, ELISA, slot blot, qPCR, or other tecnhiques, at three time points: admission and discharge from rehabilitation hospital, and follow up (one-year post-injury).

CONTACTS AND LOCATIONS:
Overall Officials: Sandra I. Vieira, Prof. Dr., Principal Investigator — Institute of Biomedicine, Department of Medical Sciences, University of Aveiro (iBiMED-UA); Maria Ribeiro da Cunha, MD, Study Director — Centro de Reabilitação do Norte (CRN)/Unidade Local de Saúde de Gaia e Espinho, E.P.E. (ULSGE)
Locations (1):
- Centro de Reabilitação do Norte (CRN) / Unidade Local de Saúde Gaia e Espinho, E.P.E. (ULSGE), Vila Nova de Gaia,, Portugal, Vila Nova de Gaia, Portugal

IPD SHARING:
Plan to Share IPD: Undecided